CLINICAL TRIAL: NCT00677521
Title: A Pilot Study of Acarbose as Treatment for Pediatric Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment and no student currently interested in working on this project.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Emeritus Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000011557
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Acarbose — 50mg tablet by mouth daily for the first 2 weeks, then twice a day for the next 2 weeks, and then three times a day for the next 8 weeks for a total of 12 weeks.

SUMMARY:
The objective of this study is to demonstrate a reduction of intrahepatic fat as measured with Proton Magnetic Resonance Spectroscopy after 12 weeks administration of oral acarbose. The study will also examine the hypothesis of whether the chronic administration of acarbose in patients with NAFLD will influence postprandial substrate metabolism reflected in the RQ measured by indirect calorimetry.

DETAILED DESCRIPTION:
The chronic administration of acarbose has been shown to improve insulin resistance and reverse impaired glucose tolerance. Both these conditions, especially insulin resistance, are physiologically associated with the development and progression of NAFLD. Therefore, we hypothesized that the chronic administration of acarbose attenuates NAFLD by improving glucose handling. This would be reflected in a reduction of intrahepatic fat accumulation. Proton Magnetic Resonance Spectroscopy is a sensitive and non-invasive method to measure changes in intrahepatic fat content. The primary endpoint of this study would be to demonstrate a reduction of intrahepatic fat as measured with Proton Magnetic Resonance Spectroscopy after 12 weeks administration of oral acarbose. Other relevant secondary outcomes that have been previously demonstrated to be associated with improvement of NAFLD included improvement of insulin resistance, normalizing of serum adiponectin, and a lowering of serum Leptin.

A second intent of the study is to test the hypothesis of whether the chronic administration of acarbose in patients with NAFLD will influence postprandial substrate metabolism reflected in the RQ measured by indirect calorimetry. The consequence of insulin resistance is a relative inhibition of fatty oxidation. However, the chronic administration of acarbose improves insulin resistance and dampens the post-prandial surge in serum glucose and insulin. These changes in glucose handling could possibly result in a shift towards a pattern of preferential lipid oxidation. We anticipate either a lowering or blunting of the postprandial RQ after chronic administration of acarbose for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age:10-18 years old
* Liver biopsy proven NAFLD. NAFLD defined histologically as greater than 5% hepatic macrovesicular steatosis with any degree of chronic inflammation and hepatic fibrosis; clinical definition requires that other liver diseases associated with fatty liver be excluded.
* Insulin resistance with HOMA-IR score >3.0
* Hepatic steatosis >5% wet weight on hepatic proton magnetic resonance spectroscopy (1H-MRS)
* INR <1.2; Conjugated Bilirubin <2umol/L and Albumin >35gm/L

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Treatment with oral hypoglycemic agents
* Ongoing participation in a formal weight loss program or interventional clinical trial
* Panhypopituitarism and genetic causes of obesity i.e. Prader-Willi syndrome
* Alcohol consumption >20 g/day
* Serum creatinine above normal range for age
* History of previous or predisposition to intestinal obstruction
* Pre-existing gastrointestinal disease i.e. inflammatory bowel disease; celiac disease
* Drugs that influence energy metabolism, intestinal transit, substrate metabolism

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Improvement of hepatic steatosis as measured by proton magnetic resonance spectroscopy | 12 weeks

SECONDARY OUTCOMES:
Postprandial substrate metabolism reflected in the respiratory quotient (RQ) measured by indirect calorimetry | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Pencharz, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada